CLINICAL TRIAL: NCT00254579
Title: A Phase 2, Open Label, Single Arm Study To Evaluate The Efficacy, Safety, Tolerability And Pharmacokinetics Of CP-675,206 In Patients With Advanced Refractory And/Or Relapsed Melanoma
Brief Title: Study of CP-675,206 in Refractory Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3671008
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Refractory Melanoma
Keywords: refractory melanoma; malignant melanoma
MeSH Terms: conditions — Melanoma | interventions — tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 15 mg/kg CP-675,206 (Experimental)
  Interventions: Drug: CP-675,206

INTERVENTIONS:
Drug: CP-675,206 — 15 mg/kg Q12W dosing regimen

SUMMARY:
CP-675,206 is a fully human monoclonal antibody (mAb). It binds to the CTLA4 molecule, which is expressed on the surface of activated T lymphocytes. CP-675,206 is thought to stimulate patients' immune systems to attack their tumors. CP-675,206 is not expected to have a direct effect on tumor cells. CP-675,206 been shown to induce durable tumor responses in patients with metastatic melanoma in Phase 1 and Phase 2 clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Surgically incurable Stage III or IV melanoma
* One prior systemic treatment for metastatic melanoma
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) PS = 0 or 1

Exclusion Criteria:

* Melanoma of ocular origin
* Received prior vaccine
* Received prior CTLA4-inhibiting agent
* History of, or significant risk for, chronic inflammatory or autoimmune disease
* Potential requirement for systemic corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2005-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To assess the anti-tumor efficacy, as determined by objective response rate, of intravenous CP-675,206 administered at a dose of 15 mg/kg every 90 days to patients with relapsed or refractory advanced melanoma | Tumor response is assessed every 2-3 months until disease progression

SECONDARY OUTCOMES:
Safety | At every scheduled visit as specified per protocol for a maximum of 2 years from first dose of drug
Pharmaco Kinetic | At every scheduled visit as specified per protocol for a maximum of 2 years from first dose of drug
Survival | At every scheduled visit as specified per protocol for a maximum of 2 years from first dose of drug
Health-related QoL | At every scheduled visit as specified per protocol for a maximum of 2 years from first dose of drug

CONTACTS AND LOCATIONS:
Locations (57):
- United States (30):
  - Research Site, Scottsdale, Arizona
  - Research Site, Bentonville, Arkansas
  - Research Site, Fayetteville, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Los Angeles, California
  - Research Site, Aurora, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Ocoee, Florida
  - Research Site, Orlando, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Durham, North Carolina
  - Pfizer Investigational Site, Columbus, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Salt Lake City, Utah
  - Research Site, Federal Way, Washington
  - Research Site, Lakewood, Washington
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Madison, Wisconsin
- Research Site, Ciudad de Buenos Aires, Buenos Aires, Argentina
- Australia (5):
  - Research Site, Waratah, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, Woolloongabba, Queensland
  - Research Site, East Melbourne, Victoria
  - Research Site, Nedlands, Western Australia
- Research Site, Hamilton, Ontario, Canada
- France (3):
  - Research Site, Lille, Cedex
  - Research Site, Paris
  - Research Site, Villejuif
- Germany (4):
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Kiel
  - Research Site, Tübingen
- Italy (2):
  - Research Site, Meldola, FC
  - Research Site, Milan
- Spain (4):
  - Research Site, Barcelona, Barcelona
  - Research Site, Madrid, Madrid
  - Research Site, Pamplona, Navarre
  - Research Site, Zaragoza, Zaragoza
- United Kingdom (7):
  - Research Site, Truro, Cornwall
  - Research Site, Northwood, Middlesex
  - Research Site, Sutton, Surrey
  - Research Site, Newcastle upon Tyne, Tyne and Wear
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne